CLINICAL TRIAL: NCT02359968
Title: PReoperative Chemoradiation With Paclitaxel-carboplatin or With Fluorouracil-oxaliplatine-acide Folinique (FOLFOX) for Resectable Esophageal and Junctional Cancer - A Randomized Phase II Trial
Brief Title: PReoperative Chemoradiation (Paclitaxel-carboplatin or FOLFOX) for Resectable Esophageal and Junctional Cancer
Acronym: PROTECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-1402
Record Dates: First submitted 2015-01-12; First posted 2015-02-10 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Neoplasms; Gastro-esophageal Junction Cancer
Keywords: resectable esophageal; junctional cancer; FOLFOX; paclitaxel-carboplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Folfox protocol; Fluorouracil; Oxaliplatin; Leucovorin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX (Active Comparator): * Fluorouracil 400 mg/m², IV bolus dose on day 1, followed by continuous IV infusion of fluorouracil 1600 mg/m² over 2 days
  * Oxaliplatin 85 mg/m², 2-hr IV infusion on day 1
  * Folinic acid 200 mg/m² 2-hr IV infusion on day 1
  * 3 cycles, q14
  Interventions: Drug: FOLFOX
- CarboP-pacliT (Experimental): * Carboplatin (carboP) AUC=2, given by intravenous infusion
  * Paclitaxel (pacliT) 50 mg/m², given by intravenous infusion
  * on days 1, 8, 15, 22 and 29
  Interventions: Drug: CarboP-pacliT

INTERVENTIONS:
Drug: FOLFOX — radiochemotherapy before surgery
  Other Names: Fluorouracil; Oxaliplatin; Folinic acid; Elvorine
  Arms: FOLFOX
Drug: CarboP-pacliT — radiochemotherapy before surgery
  Other Names: Carboplatine; paclitaxel
  Arms: CarboP-pacliT

SUMMARY:
Resectable esophageal or junctional cancer requires medical treatment by radiotherapy and chemotherapy followed by surgery. Currently, one of the most commonly used chemotherapy treatment is the FOLFOX. It is a combination of three drugs administered intravenously: fluorouracil, oxaliplatin and folinic acid. This is the standard treatment.

Another protocol of chemotherapy is widely used by certain European and American teams, due to promising results : a combination of two drugs administered intravenously: Paclitaxel and Carboplatin (CarboP-pacliT). At present, no clinical study has shown the superiority of one treatment over the other.

The objective of this Phase II study is to clarify clinical practice by comparing these two chemotherapy treatments.

DETAILED DESCRIPTION:
There is no standard preoperative (neoadjuvant) chemoradiation (NCRT) regimen for resectable esophageal cancer, because most if all trials failed to show any survival advantage favoring pCRT when compared to surgery only. This failure had been related to the lack of power of some trials, as well as the ability of chemoradiation to potentiate post-operative morbidity (including mortality), and therefore hampering the accrual of its own survival benefit. Hopefully, meta-analyses showed that NCRT increases survival when compared to surgery only. However, in the clinical practice, this does not make easier the choice of the best NCRT treatment. It appeared that the radiation regimen that were used in each randomized trials were heterogeneous with respect with dose, fraction, length of treatment, fields, dosimetry planning, and quality control. This applies also to chemotherapy with respect with the kind of cytotoxics that were used (including number of drugs), as well as dosage, and the number of cycles, although most of the time cytotoxics were fluorouracil and cisplatin.

Dutch colleagues recently showed that NCRT with weekly carboplatin and paclitaxel increase survival, without increasing postoperative mortality. Of note, most tumors in this trial arose from the lower third of the esophagus and esogastric junction and these habitually correlate with less postoperative morbidity compared to upper third tumors. Moreover, the lung volume spared from radiation was greater in junctional tumors than in upper third cancers - a critical point in the development of radiation-induced pneumonitis and subsequent postoperative mortality. It is difficult to understand how this taxane-based chemotherapy is active, as it did not make better that fluorouracil-based regimen in non-operable patients, and as NCRT with taxanes makes radiation-induced pneumonitis more likely. The favorable impact of this NCRT may lie on its radiation regimen. A moderate total dose of radiation, smaller radial margins than in other trials and modern dosimetry with 3D-planning all improve the safety of treatment and of subsequent surgery. Finally, the favorable impact of the Dutch NCRT regimen may lies on the fact that it does not include cisplatin, a compound which has been found related to the occurrence of more sudden deaths than a non cisplatin-based regimen such as the FOLFOX combination (fluorouracil, oxaliplatin, folinic acid) in the setting of definitive chemoradiotherapy.

Our aim is to evaluate the short-term benefit (complete resection rate) and safety (severe postoperative rate) of 2 preoperative regimen, (carboplatin-paclitaxel or fluorouracil-oxaliplatin-folinic acid), combined to the Dutch radiation backbone, in operable esophageal and junctional (Siewert I-II) cancer. The present trial offers the unique opportunity to compare two therapeutic strategies that have already been shown to be efficient in large randomized controlled trials offering level-1 evidence.

ELIGIBILITY:
Inclusion Criteria:

* Resectable and operable esophageal cancer located under the carena (beyond 25 cm from the incisors) or junctional cancer (Siewert I or II)
* Invasive adenocarcinoma or squamous cell type (to stick to the population included in the CROSS trial)
* Patient who present with:

  * stage IIA (T3N0M0)
  * stage IIB (T1 N1 M0 or T2 N1 M0),
  * stage III (T3 N1 M0 or T4 N0 N1 M0) tumors
* ECOG performance status 0, 1 or 2
* Patient eligible for preoperative chemoradiation with either fluorouracil- oxaliplatin-folinic acid, or Paclitaxel-carboplatin
* Age ≥ 18
* Peripheral neuropathy ≤ NCI-CTC grade 1
* Adequate bone marrow reserve, normal renal and liver functions:

  * Neutrophil count ≥ 1500/mm3
  * Platelet count ≥ 100 000/mm3
  * Hemoglobin ≥ 10 g/dl (after transfusion, if necessary)
  * Creatinin < 15mg/L
  * Clearance of creatinin (Cockcroft formulae) ≥ 60 ml/mn
  * Prothrombin time ≥ 60%
  * ASAT-ALAT ≤2.5 x ULN
  * Total bilirubin < 1.5 x ULN
  * Albumin greater the lower limit of normal
* Start of treatment within 28 days after randomization
* Negative pregnancy test (serum beta-HCG) performed within 1 week prior to start of study treatment in females with reproductive potential
* Patient covered by government health insurance
* Patient who provide a signed written informed consent form

Exclusion Criteria:

* Patient who present with stage I or stage IIA (including T2 N0 M0) or stage IV
* Patient who present with common contraindications for surgery related to patient status
* Patient who present with common contraindications for surgery related to disease extension
* Patient who present with common contraindication to radiochemotherapy with either fluorouracile-cisplatin or with paclitaxel-carboplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Short-term benefit of 2 preoperative regimen: complete resection rate AND severe (grade ≥ 3) postoperative morbidity/mortality according to the Clavien-Dindo classification | up to 30 days after surgery
  Complete resection rate (R0, that is "complete removal of all tumor with microscopic examination of margins showing no tumor cells") AND severe (grade ≥ 3) postoperative morbidity/mortality according to the Clavien-Dindo classification. Severe postoperative complication is defined by grade ≥III per-operative or post-operative complication occurring in the 30 days after surgery.

SECONDARY OUTCOMES:
Rate of completion of full treatment without modification | up to 58 days
Evaluation of the efficacy of both regimen in term of overall survival | From date of inclusion until the date of death from any cause assessed up to 36 months after the last surgery
  Overall survival using Kaplan-Meier method
Evaluation of the efficacy of both regimen in term of disease-free survival | From date of inclusion until the date of first documented progression whichever came first, assessed up to 36 months after the last surgery
  Disease-free survival using Kaplan-Meier method
Evaluation of the safety of the evaluated regimens in terms of preoperative mortality. | From registration to surgery
  Preoperative mortality (grade 5) rate, according to NCI-CTCAE v4.0 criteria
Evaluation of the safety of the evaluated regimens in terms of preoperative morbidities, postoperative morbidities, respiratory morbidities. | From start of treatment to end of study
  Pre-operative morbidities according to NCI-CTCAE v4.0 criteria, post-operative morbidities occurring in the 30 days after surgery with the main post-operative complication graded according to Clavien-Dindo, post-operative morbidities occurring more than 30 days after surgery graded according to NCI-CTCAE V4.0, postoperative respiratory morbidity rate according to the Clavien-Dindo classification.
Evaluation of the efficacy of both regimen in term of Pathological response rate | Surgery
  Complete pathological response (ypCR) rate
Evaluation of the efficacy of both regimen in term of quality of life | Up to 3 years after surgery
  Quality of life: QLQC30 and OES18

OTHER OUTCOMES:
DVH (CoDose-Volume-Histogram (DVH) and postoperative respiratory morbidity | up to 30 days after the beginning of radiotherapy
Comparison of both arms in terms of safety and efficacy | From date of inclusion until the date of death from any cause assessed up to 36 months after the last surgery
  Evaluation of preoperative mortality (grade 5) rate according to NCI-CTCAE v4.0 criteria, pre-operative morbidities according to NCI-CTCAE v4.0 criteria, post-operative morbidities occurring in the 30 days after surgery with the main post-operative complication graded according to Clavien-Dindo, post-operative morbidities occurring more than 30 days after surgery graded according to NCI-CTCAE V4.0, postoperative respiratory morbidity rate according to the Clavien-Dindo classification.
  Evaluation of overall survival and disease-free survivalusing Kaplan-Meier method, complete pathological response (ypCR) rate
Net treatment benefit estimation | From date of inclusion until the date of death from any cause assessed up to 36 months after the last surgery
  To estimate the net treatment benefit, combining efficacy and safety endpoints, using the Generalized Pairwise Comparisons Method - GPC method (Buyse, 2010)
Prognostic factor and treatment effect controlling for possible confounding factors | From date of inclusion until the date of first documented progression whichever came first, assessed up to 36 months after the last surgery
  To identify prognostic factors associated to disease-free survival, and evaluate the treatment effect controlling for possible confounding factors. Following factors will be studied: pre-therapeutic stage (II versus III), pre-therapeutic N (positive versus negative), post-surgery stage (ypT0N0 versus other), TRG (1-2 versus other) and resection (R0 versus other).

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, Principal Investigator — Centre Oscar Lambret; Guillaume PIESSEN, MD, Principal Investigator — University Hospital of Lille
Locations (10):
- France (10):
  - ICO Paul Papin, Angers
  - CHU Bordeaux, Bordeaux
  - University Hospital of Lille, Lille
  - Centre Oscar Lambret, Lille
  - Hôpital La Timone, Marseille
  - Hôpital Nord, Marseille
  - ICM - Val d'Aurelle, Montpellier
  - CH Lyon sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - ICO René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messager M, Mirabel X, Tresch E, Paumier A, Vendrely V, Dahan L, Glehen O, Vasseur F, Lacornerie T, Piessen G, El Hajbi F, Robb WB, Clisant S, Kramar A, Mariette C, Adenis A. Preoperative chemoradiation with paclitaxel-carboplatin or with fluorouracil-oxaliplatin-folinic acid (FOLFOX) for resectable esophageal and junctional cancer: the PROTECT-1402, randomized phase 2 trial. BMC Cancer. 2016 May 18;16:318. doi: 10.1186/s12885-016-2335-9. PMID 27194176